CLINICAL TRIAL: NCT05493969
Title: A Study Evaluating the Efficacy and Tolerability of Dolutegravir Plus Lamivudine in HIV Infected Adults Who Are Virologically Suppressed and With Evidence of TDF Toxicity
Brief Title: Efficacy and Tolerability of DTG Plus 3TC in HIV Infected Adults With Virologically Suppression and TDF Toxicity
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Renfang Zhang, Clinical professor, Shanghai Public Health Clinical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2432
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DTG/3TC (Other): Subjects will switch to dolutegravir (DTG) plus lamivudine (3TC) or fixed dose combination DTG/3TC for 48 weeks.
  Interventions: Drug: Dolutegravir 50 MG plus lamivudine 300 MG； Dolutegravir/lamivudine (50 MG/300 MG)

INTERVENTIONS:
Drug: Dolutegravir 50 MG plus lamivudine 300 MG； Dolutegravir/lamivudine (50 MG/300 MG) — Subjects will discontinue their TDF + 3TC/FTC-based regimen and will switch to DTG+3TC or fixed dose combination DTG/3TC.

SUMMARY:
To investigate the efficacy and tolerability of the regimen of dolutegravir plus lamivudine in HIV infected adults who are virologically suppressed and with evidence of TDF toxicity.

DETAILED DESCRIPTION:
This study is a single-center, prospective, uncontrolled, open-label and single-arm interventional study, and aim to investigate the efficacy and safety of dolutegravir plus lamivudine (DTG+3TC) for HIV-infected adults switching from TDF-based triple ART due to TDF toxicity. The study populations are : HIV-infected patients, irrespective of gender, aged 18-75 years old; At least one plasma HIV-1 RNA<40 c/mL in the 6 months prior to Screening and plasma HIV-1 RNA <40 c/mL at Screening; Must be on uninterrupted TDF + 3TC / FTC-based regimen for ≥ 6 months prior to Screening; There are clinical manifestations of TDF related adverse reactions. All enrolled subjects will receive DTG + 3TC once daily (DTG + 3TC) for up to 48 weeks. After stable switch indication approved in China mainland, it's allowed for subjects switch from DTG+3TC to fixed dose combination DTG/3TC. The primary endpoint is the percentage of participants with virologic failure at 48 weeks of treatment by FDA Snapshot algorithm. The secondary endpoints are immunologic outcomes and adverse events including bone and renal biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects were required to meet one of the following criteria: 1) Incapacitated, defined as postmenopausal (spontaneous amenorrhea at 12 months, age ≥45 years) or physically unable to conceive after tubal ligation, hysterectomy, or bilateral oophorectomy; 2) Have potential to have children, but are negative at screening and on day 1 pregnancy test, and agree to use appropriate contraceptive methods, including oral contraceptives, condoms and intrauterine devices;
2. At least once plasma HIV-1 RNA<40 c/mL in the 6 months prior to screening and plasma HIV-1 RNA <40 c/mL at screening;
3. Must be on uninterrupted TDF + 3TC/FTC-based regimen for ≥6 months prior to screening;
4. Participants with pre-existing clinical manifestations of TDF related adverse reactions at the time of screening.

   TDF-related renal damage was defined as: meeting 1 of the 5 following conditions in the investigator's judgement, based upon the medical history and relevant examinations, likely to represent TDF toxicity:

   i. eGFR decrease by 5 mL/min per year for at least 3 consecutive years or confirmed 25% eGFR decline from baseline ii. Urine β2-microglobulin/Cr ≥300 μg/g iii. Urine microalbumin/creatinine >30 μg/mg iv. Non-diabetic glycosuria (urine glucose 1+ or above) v. Serum phosphate <0.8 mmol/L TDF - associated bone toxicity is defined as a T-value less than -1.0 or Z- value less than -2.0 or fragility fracture after TDF/XTC use and other factors is excluded according to the medical history and relevant examination.
5. Sign the informed consent and be able to visit regularly according to the test requirements.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding or plan to become pregnant or breastfeed during the study;
2. Participants with AIDS-related opportunistic infections or AIDS-related or unrelated neoplastic diseases;
3. Patients with ALT >= 5 x ULN, or ALT >=3 x ULN and bilirubin >= 1.5xULN (with >35% direct bilirubin. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
4. Evidence of Hepatitis B virus (HBV) infection: Participants positive for HBsAg, negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded.
5. Hepatitis C virus (HCV) infection;
6. Participants who are allergic or intolerant to lamivudine or dolutegravir;
7. Participants with known previous episodes of virologic failure and known resistance mutations of 3TC or INSTI if resistance mutations had previously been identified;
8. Taking medications that contraindicated with lamivudine or dolutegravir; Other conditions that the investigator considers unsuitable to participate in the study, including the risk of suicide, poor adherence, and interference with the evaluation of clinical study endpoints.
9. Participants with creatinine clearance <30ml/min.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Virologic outcomes | Week 48
  Percentage of participants with virologic failure after 48 weeks of treatment by FDA Snapshot algorithm.

SECONDARY OUTCOMES:
HIV-RNA | Week 24 and Week 48
  Percentage of participants with HIV-RNA <40 copies/mL at weeks 24 and 48
CD4 counts | Week 24 and Week 48
  Changes from Baseline in CD4+ Cell Counts at Week 24 and 48
bone markers | Week 48
  Median percentage improvement (±SD) of circulating bone markers (alkaline phosphatase, osteocalcin, 25-OH-vitamin D level) at 24 weeks and 48 weeks after switch vs baseline)
DEXA | Week 48
  Percentage change of T-score classification (normal, osteopenia and osteoporosis) or Z-score classification (normal, abnormal) of bone mineral density using DEXA at 48 weeks after switch vs baseline
renal markers | Week 24 and Week 48
  Median percentage improvement (±SD) of urine microalbumin , serum CysC, urine β2-microglobulin/creatinine, urine N-Acetyl-Beta-D-Glucosaminidase (NAG), serum retinol binding protein (RBP) at 24 weeks and 48 weeks after switch vs baseline
eGFR | Week 24 and Week 48
  Median percentage improvement (±SD) of eGFR and Percentage change of renal function (normal, mild, moderate and severe) at 24 weeks and 48 weeks after switch vs baseline

CONTACTS AND LOCATIONS:
Overall Officials: Renfang Zhang, Study Chair — Shanghai Public Health Clinical Center

IPD SHARING:
Plan to Share IPD: No